CLINICAL TRIAL: NCT07342855
Title: Comparison Study to Evaluate the Outcomes Among Children Participating in a Community Healthy Lifestyle Program
Brief Title: Comparing Outcomes Among Children With Obesity in a Community Healthy Lifestyle Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Principal Investigator, Sarah Barlow, Professor of Pediatrics, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 73357
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Obesity; Pediatric Overweight; Overweight , Obesity
Keywords: Obesity; FNPA; BAQ; Endurance; %BMIp95; Family Healthy Weight Program; Community Healthy Lifestyle Program; intensive health behavior and lifestyle treatment; PACER
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Control group procedures The wait list control subjects will receive no intervention for 3 months. They will undergo a Time 2 measure and then begin participation in the session at the subsequent quarter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program Intervention Arm (Experimental): Participation in Get Up & Go Healthy Lifestyle Program
  Interventions: Behavioral: Get Up & Go Healthy Lifestyle Program
- Waitlist Control Arm (No Intervention): Waitlist control patients will participate in the program 3 months later

INTERVENTIONS:
Behavioral: Get Up & Go Healthy Lifestyle Program — This study evaluates an established pediatric healthy weight program, Get Up & Go. There are 10 weekly sessions for child (ages 6-14 years) and parent. Each 90-minutes session includes an interactive lesson on some aspect of healthy living, a fun game or physical activity that involves both children and parents, a healthy snack, and a time for families to set a lifestyle change goal for the week and to review achievement of goals set the prior week. Virtual components bring the total content exposure to over 26 hours provided.
  Curriculum:
  Principles of healthy living Healthy eating basics Division of responsibility Nutrition 101 Bullying prevention Meal time Advertising and dining Grocery store tour Graduation
  Arms: Program Intervention Arm

SUMMARY:
This study aims to evaluate the outcomes of an existing clinical program that teaches families of children with overweight and obesity healthy lifestyle. The design will be unblinded, randomized, waitlist control.

DETAILED DESCRIPTION:
The participants will come from the cohort of patients who are referred to the Get Up & Go program and decide to enroll. For this existing family healthy weight program, the child must be between 6 and 14 years of age at time of program start, with BMI by report of ≥ 85th percentile. The child must be able to participate in physical activity comparable to an elementary school PE class and must be able to function cognitively at or above the level of a 6 year old.

The process for enrollment in this program begins with a standard referral that goes to the Get Up & Go office at Children's Health. Staff will make referred families aware of study at initial contact; staff generally place a call to families to give overview of Get Up & Go. Office staff tell interested families that they will be contacted closer to the time of class start. Whether or not the family answers the phone, the family is mailed a welcome packet.

For the study, the Get Up & Go staff will inform families by phone that they may qualify for a study that performs additional measures to help understand the effect of the program. These families will hear that study participation is optional. The staff will tell the families that a study coordinator will call or text unless the family says they do not want to be contacted. The welcome packet will include a page with the same information and an opt-out postcard. To enroll in this study, the parent must speak English or Spanish.

The study coordinator will call families who have not declined contact, up to 5 times at different times of day. When they reach the family, they will review the study protocol and invite participation. The coordinator will review the study protocol, explaining that participation will mean a 1-hour visit measure several weeks prior to class start and agreement to accept randomization to immediate start or 3 months deferment. If family wants to enroll, the consent will be reviewed, and all questions answered. The parent will verbally consent and will receive a copy of the (unsigned per IRB waiver) consent via email. The child will assent. If families prefer, they can defer consent or assent until the in-person appointment for measurement.

A study coordinator will schedule a time 1-4 weeks before the start of the Get Up & Go class to meet with a small group (1-5) of study families at either the YMCA or at Children's Health to perform baseline measures. If any families were interested but did not consent virtually, they will undergo consenting process at this time. When measures (see description below) are complete, a simple 1:1 randomization will be done, using a computer software program that generates random sequence. Neither research team nor family will be blinded to assignment

1. Intervention: immediate participation
2. Control: Waitlist, deferring participation for approximately 3 months, to the next quarter

The wait list control subjects will receive no intervention for 3 months. They will undergo a Time 2 measure and then begin participation in the session at the subsequent quarter.

Data collected will include height, weight, %BMIp95, endurance via PACER test. Survey data: The Family and Nutrition and Physical Activity (FNPA) and Behavior Assessment Questionnaire (BAQ).

Optional data: Parental height, weight, and BMI.

Each quarter, approximately 40 families will be enrolled, with 20 randomized to start immediately and 20 to wait until the subsequent quarter. Cohorts will be recruited each quarter for 4-5 quarters until enrollment is complete.

ELIGIBILITY:
Inclusion Criteria:

* BMI by report of ≥ 85th percentile
* The child must be able to participate in physical activity comparable to an elementary school PE class and must be able to function cognitively at or above the level of a 6 year old

Exclusion Criteria:

* BMI by report of below the 85th percentile
* Inability to participate in physical activity comparable to an elementary school PE class and must be able to function cognitively at or above the level of a 6 year old

Parent will be invited but not required to be weighed and measured.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
BMI status | From enrollment to the end of intervention period at 3 months
  Change in child BMI status, using %BMIp95 as primary outcome and BMI z score. Both are calculations made from weight, height, sex, and age.

SECONDARY OUTCOMES:
Family Nutrition and Physical Activity (FNPA) | From enrollment to the end of intervention period at 3 months
  Family Nutrition and Physical Activity (FNPA), a validated 30-item questionnaire from the Academy of Nutrition and Dietetics, will be completed by parent.
  The questions ask about home practices related to nutrition, physical activity, sleep and other health routines. The instrument has been broadly utilized since it was validated in 2009 . The FNPA has been used to assess modifiable healthy lifestyle behaviors, with an emphasis on behaviors that contribute to obesity .
  Each questions are rated on a scale of 1 to 4. Higher aggregate scores point to healthier decision making. Lower scores point to less healthy behaviors.
BAQ: Behavior Assessment Questionnaire | From enrollment to the end of intervention period at 3 months
  Behavior Assessment Questionnaire (BAQ) is a self reported tool measuring a child's lifestyle behaviors. It examines frequency of habits such as eating, activity, emotional health, sleep, and environment. Each of the 10 questions has 4 response options describing frequency or timing of stem question. The responses are assigned scores of 0-4, and total scores are converted to a 0-100 scale. Higher aggregate scores point to healthier habits, and lower scores point to less healthy behaviors.
Endurance (PACER) | From enrollment to the end of intervention period at 3 months
  Progressive Aerobic Cardiovascular Endurance Run (PACER): participants run a 15 m distance at a progressively faster pace, and the score is the number of laps successfully completed
Parental Weight Measures | From enrollment to the end of intervention period at 3 months
  Optional: Parent BMI, using absolute BMI (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern, Children's Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient BMI changes, pacer results, questionnaire results.
Supporting Information: Study Protocol, CSR
Time Frame: Deidentified IPD underlying the results reported for the study can be available beginning 6 months after publication and ending 3 years after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data will can be sent via a secure method.

REFERENCES:
- [Background] O'Connor EA, Evans CV, Henninger M, Redmond N, Senger CA. Interventions for Weight Management in Children and Adolescents: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2024 Jul 16;332(3):233-248. doi: 10.1001/jama.2024.6739. PMID 38888913
- [Background] O'Connor EA, Evans CV, Burda BU, Walsh ES, Eder M, Lozano P. Screening for Obesity and Intervention for Weight Management in Children and Adolescents: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2017 Jun 20;317(23):2427-2444. doi: 10.1001/jama.2017.0332. PMID 28632873
- [Background] Barlow SE, Lorenzi A, Reid A, Huang R, Yudkin JS, Messiah SE. The Implementation and Five-Year Evolution of a Childhood Healthy Weight Program: Making a Health Care-Community Partnership Work. Child Obes. 2021 Oct;17(7):432-441. doi: 10.1089/chi.2021.0010. Epub 2021 May 3. PMID 33945306
- [Background] Chiong R, Gray VB, Roy R. Development of a Family-Based Nutrition Program Rooted in Food Parenting Literature. Fam Consum Sci Res J. 2020 Sep;49(1):67-83. Epub 2020 Aug 28. PMID 33239856
- [Background] Yudkin JS, Allicock MA, Atem FD, Galeener CA, Messiah SE, Barlow SE. Efficacy of a Primary Care eHealth Obesity Treatment Pilot Intervention Developed for Vulnerable Pediatric Patients. Child Obes. 2024 Mar;20(2):75-86. doi: 10.1089/chi.2022.0185. Epub 2023 Mar 9. PMID 36893214
- [Background] Ihmels MA, Welk GJ, Eisenmann JC, Nusser SM. Development and preliminary validation of a Family Nutrition and Physical Activity (FNPA) screening tool. Int J Behav Nutr Phys Act. 2009 Mar 12;6:14. doi: 10.1186/1479-5868-6-14. PMID 19284631
- See also: Get Up & Go Website — https://www.childrens.com/specialties-services/specialty-centers-and-programs/endocrinology/programs-and-services/get-up-and-go